CLINICAL TRIAL: NCT03626064
Title: Management and Point-of-Care for Tobacco Dependence (PROMPT): a Feasibility Mixed Methods Community-based Participatory Action Research Project in Ottawa, Canada
Brief Title: The PROMPT Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20140333-01H
Record Dates: First submitted 2018-06-11; First posted 2018-08-10 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2018-08

CONDITIONS: Tobacco Use Disorder; Tobacco Dependence; Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PROMPT Participants (Other): 80 participants who are homeless or at-risk for homelessness, smoke tobacco, and identify as People Who Use Drugs in Ottawa.
  Interventions: Behavioral: Smoking Cessation Counselling; Drug: Nicotine Replacement Therapy

INTERVENTIONS:
Behavioral: Smoking Cessation Counselling — One on one smoking cessation counselling with a certified mental health nurse
Drug: Nicotine Replacement Therapy — Access to a range of nicotine replacement therapy: nicotine patch, nicotine gum, nicotine lozenge, nicotine inhaler

SUMMARY:
The PROMPT Pilot Study is a feasibility mixed methods prospective cohort study following principles of community-based participatory action research. The study recruited 80 people who use drugs and followed them for 6 months while providing access to counselling, nicotine replacement therapy and peer-support in a community setting. A notable reduction in average cigarette use per day (20.5 to 9.3) and illicit substance use (18.8%) was observed at study-end. PROMPT's patient engagement model is an effective harm-reduction strategy for the growing opioid use crisis and can improve the health outcomes of marginalised at-risk populations worldwide.

DETAILED DESCRIPTION:
Objective To determine the feasibility of a Community-Based Participatory Tobacco Dependence Strategy (PROMPT) in the inner city population of Ottawa (Canada).

Design A feasibility mixed methods prospective cohort study following principles of community-based participatory action research.

Intervention Recruited 80 people who use drugs, followed them for 6 months while providing access to counseling, nicotine replacement therapy and peer-support in a community setting.

Setting Community research office in downtown Ottawa, adjacent to low-income housing, shelter services and street-based drug consumption.

Primary outcome Retention rate at 6-month follow-up.

Secondary outcome Biochemically validated 7-day point prevalence smoking abstinence at 26 weeks, self-reported abstinence in the past 7 days with exhaled carbon monoxide ≤10 ppm.

ELIGIBILITY:
Inclusion Criteria:

* currently living in Ottawa for at least 3 months prior to enrolment
* 16 years or older
* have used drugs in the past year (excluding marijuana and alcohol)
* have smoked tobacco in the past 7 days

Exclusion Criteria:

* consent declined (refusal from participant or decision maker)
* any person accessing addictions treatment (in-patient drug rehabilitation) and hence unavailable for follow-up
* any person currently or recently (in the past 30 days) enrolled in a smoking cessation program
* anyone with a terminal illness with a life expectancy of <3 months.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Retention of Study Participants | 6 months
  Retention rate at 6-month follow-up

SECONDARY OUTCOMES:
Biochemical Validation of Smoking Cessation Outcome | 6 months
  Biochemically validated 7-day point prevalence smoking abstinence at 26 weeks, self-reported abstinence in the past 7 days with exhaled carbon monoxide ≤10 ppm.

IPD SHARING:
Plan to Share IPD: Yes
Data will be available to researchers that contact the Principal Investigator.
Supporting Information: SAP
Time Frame: Data will be available upon request for the period decided necessary by the Principal Investigator and the inquiring researcher or researchers.
Access Criteria: Will provide access in the manner decided by Principal Investigator and the inquiring researcher or researchers.

REFERENCES:
- [Derived] Pakhale S, Visentin C, Tariq S, Kaur T, Florence K, Bignell T, Jama S, Huynh N, Boyd R, Haddad J, Alvarez GG. Lung disease burden assessment by oscillometry in a systematically disadvantaged urban population experiencing homelessness or at-risk for homelessness in Ottawa, Canada from a prospective observational study. BMC Pulm Med. 2022 Jun 16;22(1):235. doi: 10.1186/s12890-022-02030-x. PMID 35710334
- [Derived] Pakhale S, Tariq S, Huynh N, Jama S, Kaur T, Charron C, Florence K, Nur F, Bustamante-Bawagan ME, Bignell T, Boyd R, Haddad J, Kendzerska T, Alvarez G. Prevalence and burden of obstructive lung disease in the urban poor population of Ottawa, Canada: a community-based mixed-method, observational study. BMC Public Health. 2021 Jan 21;21(1):183. doi: 10.1186/s12889-021-10209-w. PMID 33478466